CLINICAL TRIAL: NCT01961063
Title: Safety and Feasibility of Gene Transfer After Frontline Chemotherapy for Non-Hodgkin Lymphoma in AIDS Patients Using Peripheral Blood Stem/Progenitor Cells Treated With a Lentivirus Vector-Encoding Multiple Anti-HIV RNAs
Brief Title: Gene Therapy After Frontline Chemotherapy in Treating Patients With AIDS-Related Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13282; NCI-2013-01728 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13282 (Other: City of Hope Medical Center)
Record Dates: First submitted 2013-09-09; First posted 2013-10-11 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: AIDS-related Non-Hodgkin Lymphoma; AIDS-related Plasmablastic Lymphoma; AIDS-related Primary Effusion Lymphoma; HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (gene therapy) (Experimental): Patients receive busulfan IV over 3 hours on day -2 followed by lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells IV on day 0.
  Interventions: Drug: busulfan; Biological: lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: busulfan — Given IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Biological: lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells — Given IV
  Other Names: lentivirus-transduced hematopoietic progenitor cells
Other: pharmacological study — Correlative studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies gene therapy after frontline chemotherapy in treating patients with acquired immune deficiency syndrome (AIDS)-related non-Hodgkin lymphoma (NHL). Placing genes for anti-human immunodeficiency virus (HIV) ribonucleic acid (RNA) into stem/progenitor cells may make the body build an immune response to AIDS. Giving the chemotherapy drug busulfan before gene therapy can help gene-modified cells engraft and work better.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and feasibility of recombinant (r)HIV7-short hairpin RNA targeted to the HIV-1 tat/rev (shI)-trans-active response element (TAR)-chemokine cysteine-cysteine receptor 5 ribozyme (CCR5RZ)-treated hematopoietic stem progenitor cells (HSPC) (lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells) infusion in AIDS patients completing treatment for NHL and non-myeloablative conditioning with busulfan.

II. To demonstrate the engraftment of gene-modified progeny cells following such treatment.

III. To determine if selection of these gene-modified progeny cells occurs during analytical treatment interruption (ATI) of combination anti-retroviral therapy (cART).

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of busulfan in patients with AIDS-related lymphoma (ARL).

II. To determine the effects of HIV-1 infection on the presence of gene-marked peripheral blood mononuclear cells (PBMC) as measured by woodchuck post-transcriptional regulatory element (WPRE) deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) performed before, during, and after ATI.

OUTLINE: Patients receive busulfan intravenously (IV) over 3 hours on day -2 followed by lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells IV on day 0.

After completion of study treatment, patients are followed up at 1, 7, 14, and 21 days and 1, 2, 3, 6, 9, 12, 18, and 24 months and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive at or before the time of lymphoma diagnosis
* Karnofsky performance status >= 70%
* Biopsy proven NHL, including plasmablastic lymphoma and primary effusion lymphoma but not T-cell lymphoma; tissue histology will be reviewed at City of Hope (COH); patients who have been in remission for > 1 year post Hodgkin's lymphoma chemotherapy are also considered eligible
* >= 28 days from completion of frontline chemotherapy for NHL
* If remission status < 1 year for NHL, complete remission documented by computed tomography (CT) or positron emission tomography (PET)-CT scan within 3 months of study entry
* No diagnosed psychosocial conditions that would hinder study compliance and follow-up
* Pretreatment serum glutamic oxaloacetic transaminase (SGOT), serum glutamate pyruvate transaminase (SGPT) =< 2.5 x institutional upper limit of normal (ULN)
* Pretreatment serum bilirubin =< 2.5 x institutional ULN or - Total bilirubin < 4.5 mg/dl with direct fraction =< 0.3 mg/dl in patients for whom these abnormalities are felt to be due to protease inhibitor therapy
* Serum creatinine < 2 x the institutional ULN
* Absence of clinically significant cardiomyopathy, congestive heart failure
* Cardiac ejection fraction has to be >= 50%
* Spirometry diffusion capacity (diffusion capacity of the lung for carbon monoxide [DLCO]) >= 50%
* If the subject is female and of child-bearing potential, subject must have negative serum or urine pregnancy test within 7 days of treatment with research agent; men with partners of child-bearing potential and women of child-bearing potential must be willing to use medically effective birth control methods, e.g. contraceptive pill, condom, or diaphragm and continue this for one year post HSPC infusion
* Subjects must be on a prophylactic regimen for Pneumocystis carinii pneumonia, or agree to begin such treatment, if the cluster of differentiation (CD)4 counts are < 200 cells/uL

SECONDARY ELIGIBILITY CRITERIA FOR GENE-MODIFIED HSPC INFUSION:

* Subjects must complete the filgrastim (G-CSF)/plerixafor mobilization of peripheral blood progenitor cells and must have collected at least 7.5 x 10^6 CD34+ cells/kg, sufficient for preparation of both, a back-up of 2.5 x 10^6 CD34+ cells and the research product
* Research product must pass all release tests
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Any AIDS-related opportunistic infection occurring within the past year and for which treatment has been unsuccessful would be considered exclusionary, but this is done on a case-by-case basis as determined by the principal investigator
* Active cytomegalovirus (CMV) retinitis or other active CMV-related organ dysfunction; patients with a history of treated CMV infection are not excluded
* Patients who are hepatitis C virus (HCV) antibody positive and HCV ribonucleic acid (RNA) or hepatitis B virus (HBV) surface antigen positive and HBV DNA positive
* Pregnant or nursing women
* Active central nervous system (CNS) lymphoma, history of HIV-associated encephalopathy; dementia of any kind; seizures in the past 12 months; patients with a history of positive cerebrospinal fluid cytology that has become negative with intrathecal chemotherapy and the patient has been in remission for at least 12 months are eligible
* Any history of HIV-1 associated encephalopathy; dementia of any kind; seizures in the past 12 months; any perceived inability to directly provide informed consent (note: consent may not be obtained by means of a legal guardian)
* Any medical or physical contraindication or any other inability to undergo HSPC collection
* Patients should not have any uncontrolled illness including ongoing or active infection
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to G-CSF/filgrastim (Escherichia [E] coli producing cell line), plerixafor or busulfan
* Patients with other active malignancies other than skin cancers are ineligible for this study
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study will be considered non-compliant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2015-12-31 (Actual); Primary Completion 2026-08-05 (Estimated); Study Completion 2026-08-05 (Estimated)

PRIMARY OUTCOMES:
Procedure related toxicity as determined by adverse events (AE) grading scale using the Common Terminology Criteria for Adverse Events (CTCAE) version v4.03 | Up to 5 years
  Tables will be created to summarize these toxicities and side effects by dose
Time to Absolute Neutrophil Count (ANC) >= 500/uL | First 28 days
Time to platelet recovery to >= 50,000/uL | First 90 days

SECONDARY OUTCOMES:
Evidence for and duration of vector-marked PBMC/marrow cells assessed by PCR | Up to 5 years
  PCR-based assay on PBMC
Expression of the RNA transgenes in lineage-specific progeny of the transduced cells assessed by PCR | Up to 2 years
  PCR-based assay on FACS-sorted cells
Effect of ATI on HIV markers and CD4 count | Up to 5 years
  HIV proviral DNA, HIV RNA single copy, and 2-LTR circle DNA from PBMCs
Pharmacokinetic parameters of busulfan | Day -2 at 0 hours (pre-infusion); 3 hours (just before end of infusion); and at 4, 5, and 6 hours and day -1 at 24 hours
  Cmax, CLsys, Vd, t1/2's, AUC
Ability to obtain suitable numbers of transduced HSPC for engraftment assessed by FACS | Up to day -2 (Pre-infusion of the investigational drug)
  The number and type of cells will be determined by fluorescence activated cell sorting (FACS) analysis of the final cell product. The minimum target number of CD34+ cells for collection is 7.5 x 10e6 cells/kg and, in the final transduced cell product, the number of CD34+ cells must be >= 2.0 x 10e6 CD34+ cells/kg with total viability >= 70%.
Feasibility of product manufacturing as evidenced by product release assessed by release assays | Up to day -2 (Pre-infusion of the investigational drug)
  Release assays

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Krishnan, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States